CLINICAL TRIAL: NCT07072806
Title: Diffusion Characteristics and Efficacy of Letibotulinum Toxin A in Forehead Wrinkle Treatment
Brief Title: A Study Comparing the Safety, Efficacy, and Diffusion of Letibotulinum Toxin A Versus Other Botulinum Toxin Products in Adults With Moderate-to-Severe Forehead Wrinkles
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Collaborators: Korea International Cooperation Agency (KOICA) (Unknown)
Responsible Party: Principal Investigator, Ngoc Ha Nguyen, Dr., Yonsei University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2021-1097
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Forehead Rhytides
Keywords: Diffusion; botulinum toxin; forehead wrinkle; split-face; controlled trial
MeSH Terms: interventions — onabotulinum toxin A; Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: For each participant, the forehead was divided along the midline, with one side randomly assigned to receive the letibotulinum toxin A (Botulax®; intervention group) and the contralateral side assigned to receive one of two comparator botulinum toxin A formulations, prabotulinum toxin A (Nabota®) or onabotulinum toxin A (Botox®) (control groups 1 and 2, respectively)
Who Masked: Care Provider, Investigator
Masking Description: The allocation of treatment to the left or right side of the forehead was determined according to the randomization schedule and was concealed from both the investigators administering the treatment and the evaluators conducting outcome assessments, thereby maintaining a double-blind protocol throughout the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm A (Active Comparator): The first treatment group received letibotulinum toxin A (Botulax) on one randomly assigned side of their face and prabotulinum toxin A (Nabota) on the other side of their face.
  Interventions: Drug: Letibotulinum toxin A; Drug: Prabotulinum toxin A
- Treatment arm B (Active Comparator): The first treatment group received letibotulinum toxin A (Botulax) on one randomly assigned side of their face and onabotulinum toxin A (Botox) on the other side of their face.
  Interventions: Drug: Letibotulinum toxin A; Drug: Onabotulinum toxin A

INTERVENTIONS:
Drug: Letibotulinum toxin A — Letibotulinum toxin A (Botulax) is a botulinum toxin type A formulation developed for aesthetic indications. In this trial, it was administered as the test intervention. Each participant received 2 units injected at four forehead sites (total 8 units), diluted to 20 U/mL, on one side of the forehead. The diffusion characteristics and efficacy were compared with those of onabotulinum and prabotulinum toxin A in a double-blind, randomized, split-face design.
  Other Names: Botulax
Drug: Prabotulinum toxin A — Prabotulinum toxin A (Nabota) is a botulinum toxin type A product approved for aesthetic use in South Korea and other countries. It was used as a comparator agent in this trial. Participants received subcutaneous injections at four forehead sites (2 units per site, 8 units total), diluted to 20 U/mL, on one side of the forehead in a randomized, split-face design.
  Other Names: Nabota
  Arms: Treatment arm A
Drug: Onabotulinum toxin A — Onabotulinum toxin A (Botox) is an FDA-approved botulinum neurotoxin type A formulation used for cosmetic treatment of glabellar lines and other facial wrinkles. In this study, it was injected subcutaneously into the forehead at four standardized sites at a dose of 2 units per site (8 units total), diluted to 20 U/mL, and used as a comparator in the split-face design.
  Other Names: Botox
  Arms: Treatment arm B

SUMMARY:
The goal of this clinical trial is to learn if letibotulinum toxin A is effective and safe for treating moderate-to-severe horizontal forehead wrinkles in adults. It will also compare its diffusion characteristics with two other botulinum toxin A products. The main questions it aims to answer are:

1. Does letibotulinum toxin A reduce forehead wrinkles as effectively as other botulinum toxin A products?
2. Does letibotulinum toxin A show more localized (smaller) diffusion after injection?

Researchers will compare letibotulinum toxin A with prabotulinum toxin A and onabotulinum toxin A (Botox®) to evaluate their diffusion profiles and wrinkle-reduction effects.

Participants will:

1. Receive botulinum toxin A injections on each side of the forehead (split-face design)
2. Undergo wrinkle assessments and sweat gland function testing using 3D imaging and iodine-starch tests
3. Return to the clinic 2 weeks after treatment for follow-up evaluation

ELIGIBILITY:
Inclusion Criteria:

* Participants were eligible if they were aged ≥20 years with visible horizontal forehead wrinkles scored as moderate to severe on the Facial Wrinkle Scale using a photonumeric guide

Exclusion Criteria:

* Exclusion criteria included a history of BoNT-A injection or cosmetic procedures near the fore-head/orbital area within the past year; signs of infection or inflammation at the injection site; compen-satory frontal hyperactivity; neuromuscular disorders including myasthenia gravis or amyotrophic lateral sclerosis; use of anticoagulants, aminoglycosides, curare-like agents, or neuromuscular inhibitors (stable doses of muscle relaxants or benzodiazepines are permitted); and hypersensitivity to the inves-tigational product or iodine.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Area of Anhidrosis | 2 weeks post-injection
  The area of anhidrosis (sweat suppression) at each injection site will be measured using the Minor iodine-starch test to evaluate diffusion characteristics of botulinum toxin A formulations. The test is conducted under controlled temperature and humidity. Image-based quantification will be used to calculate the diffusion area in cm².

SECONDARY OUTCOMES:
Wrinkle Improvement | Baseline and 2 weeks post-treatment
  Wrinkle improvement was assessed 2 weeks after injection using digital photography and 3D imaging systems. Antera 3D was used to quantify the indentation index and maximal wrinkle relaxation length. Morpheus imaging was employed for three-dimensional visualization of muscle contraction and to evaluate maximal wrinkle depth. Measurements were taken on both lateral and medial sections of the forehead.

OTHER OUTCOMES:
Safety and Local Tolerability of Botulinum Toxin A Products | From baseline to 2 weeks post-injection
  All adverse events were monitored and recorded throughout the study. Severity and causal relationship to the investigational products were evaluated by the investigators. Serious adverse events were reported according to a predefined protocol. Local tolerability assessments focused on erythema, swelling, hypersensitivity reactions, and muscle weakness at injection sites.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy concerns and institutional policies that restrict data sharing beyond the research team. Data were collected under a protocol that did not include participant consent for public or external data sharing.